CLINICAL TRIAL: NCT03596970
Title: A 24-month Multi-center, Open-label, Randomized, Controlled Study to Evaluate the Evolution of Renal Function in Maintenance Liver Transplant Recipients Receiving Either RAD001 (Everolimus) Plus Reduced TAC or RAD001 (Everolimus) Plus Mycophenolate Mofetil (MMF)
Brief Title: Study of the Effect of Everolimus Immunosuppressive Combination Therapies on Renal Function When Used as a Maintenance Treatment for Liver Transplant Patients.
Acronym: Prometheus
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001HDE53
Record Dates: First submitted 2015-06-25; First posted 2018-07-24 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Liver Transplantation
Keywords: Open-label; randomized; calcineurin-inhibitor; CNI; tacrolimus; MMF; maintenance liver transplant; RAD001H; CRAD001H; liver transplant; transplantation
MeSH Terms: interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Everolimus with MMF (TAC-withdrawal) (Experimental): Everolimus (RAD001) with MMF and Steroids
  Interventions: Drug: TAC withdrawal
- Everolimus with reduced TAC (Active Comparator): Everolimus (RAD001) with reduced TAC and Steroids
  Interventions: Drug: Everolimus with reduced TAC

INTERVENTIONS:
Drug: TAC withdrawal — Everolimus (RAD001) with MMF and Steroids
  Arms: Everolimus with MMF (TAC-withdrawal)
Drug: Everolimus with reduced TAC — Active comparator arm: Everolimus (RAD001) with reduced TAC and Steroids
  Arms: Everolimus with reduced TAC

SUMMARY:
A 24-month multi-center, open-label, randomized, controlled study to evaluate the evolution of renal function in maintenance liver transplant recipients receiving everolimus plus reduced TAC or everolimus plus mycophenolate mofetil (MMF)

ELIGIBILITY:
Inclusion Criteria:

* Patients willing and capable of providing written informed consent for study participation.
* Adults 18 to 70 years of age.
* Liver allograft from a deceased or living donor.
* Treated with a CNI containing immunosuppressive regimen.
* Liver transplant 6 to 24 months prior to screening.
* Estimated kidney function between chronic kidney disease (CKD) IIIb/ 30 mL/min < eGFR < CKD II/60 mL/min with deteriorating renal function.
* Acceptable graft function (according to liver enzymes (AST / ALT) and total bilirubin).

Exclusion Criteria:

* Multiple solid organ transplant recipients
* Active chronic inflammatory bowel disease and recurrent autoimmune hepatitis
* Malignant diseases other than neoplasms of the skin.
* Patient on other investigational drug or presence of any hypersensitivity to the interventional drug.
* Pregnant or nursing (lactating) women.
* Women of child-bearing potential (physiologically capable of becoming pregnant, unless they are using effective methods of contraception).
* Anemia, thrombocytopenia, leucopenia, uncontrolled hyperlipidemia or proteinuria
* HIV positivity

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Renal Function | Randomization to Month 6
  The primary variable will be the mean change in renal function assessed by eGFR from randomization to Month 6.

SECONDARY OUTCOMES:
Efficacy (tBPAR, graft loss, death, loss to follow-up) | To Month 6
  Composite efficacy failure of tBPAR, graft loss, death or loss to follow-up and each of its components at month 6 will be analysed per event rate estimates, Kaplan-Meier and regression models. The time to the first occurrence of the event will be calculated from the randomization date.

OTHER OUTCOMES:
Number of participants with adverse events | at 24 months (end of study)
  Routine safety will be assessed via AE reporting, vital signs, and laboratory data.